CLINICAL TRIAL: NCT06078189
Title: Comparing Short-Term Functional Recovery After Surgery for Rhizarthrosis: Arthroplasty vs. Trapezectomy - A Prospective Randomized Evaluation
Brief Title: Rhizarthrosis Surgery and Functional Recovery: Arthroplasty vs. Trapezectomy
Acronym: TRAPEzE
Status: Recruiting | Type: Observational
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02775-38
Record Dates: First submitted 2023-04-11; First posted 2023-10-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Rhizarthrosis
Keywords: osteoarthritis - Trapezectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Trapezectomy group
- Experimental: Arthroplasty group
  Interventions: Device: HORUS

INTERVENTIONS:
Device: HORUS — The trapezium-metacarpal arthroplasty consists of the installation of a bipolar prosthesis composed of a metacarpal implant and a trapezial implant articulated through a metacarpal "head".
  Groups: Experimental

SUMMARY:
Rhizarthrosis is a form of osteoarthritis that affects the trapeziometacarpal joint at the base of the thumb, which is more common in women over 50. Genetic and hormonal factors as well as the frequency of certain physical movements may contribute to its appearance. Surgical treatment is recommended if medical treatment fails, and trapezectomy is currently considered the standard method, although 3rd generation trapeziometacarpal prostheses are also available.

The aim of this study is to compare the clinical and radiographic results after surgical treatment of rhizarthrosis: prosthesis versus trapezectomy.

DETAILED DESCRIPTION:
This is a two-center, randomized, prospective, comparative study.

The functional, clinical and radiographic evaluation in the early, medium and long term will make it possible to determine the possible superiority of arthroplasty if it exists.

The close evaluation of the patients during the first 3 months will make it possible to update the superiority of the arthroplasty on the functional recovery in the short term if it exists.

ELIGIBILITY:
Inclusion Criteria:

1. Age >45 years
2. Symptomatic trapezius-metacarpal osteoarthritis after failure of medical treatment ( night orthosis 3 months + failure of 2 infiltrations/year)
3. Patient who has given his/her consent to participate in the study after being informed by the surgeon,
4. Patient living in France and able to answer the survey alone.
5. Subject affiliated to a social security system or beneficiary of such a system
6. No participation in any other clinical study

Exclusion Criteria:

1. Minor patient
2. Trapezium height < 8 mm
3. Major subject protected by law, under curatorship or guardianship
4. Known allergy to the materials of the medical device
5. Local infection
6. Local skin necrosis or unhealed wound
7. Pregnant or nursing women

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic disabling osteoarthritis in failure of medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
patient assessment of the wrist | 4 weeks
  Quick-Dash score (11 minimum value and 55 is maximum
  )

SECONDARY OUTCOMES:
patient assessment of the wrist pain | 4 weeks
  Visual Analogical Assessment score (0 no pain 10 severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique BIZET, Paris, France